CLINICAL TRIAL: NCT06556108
Title: A Single-Arm, Single-Center, Open-Label Pilot Study of Anti-ALPP CAR-T Cells for Alkaline Phosphatase, Placental (ALPP)-Positive Advanced Solid Tumors
Brief Title: ALPP CAR-T Cells for ALPP-Positive Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Qingzhu Jia, M.D., Director, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQDC20191101
Record Dates: First submitted 2022-02-10; First posted 2024-08-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): This clinical study consists of 4 dose groups, with dose groups 1 and 2 using an accelerated titration dose escalation method, and dose groups 3 and 4 using a "3+3" dose escalation method.
  Interventions:
  Biological: CAR-T cells Drug: Fludarabine Drug: Cyclophosphamide
  Interventions: Biological: ALPP CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: ALPP CAR-T cells — T cells genetically engineered with a CAR targeting ALPP (ALPP CAR) that display specific reactivity against ALPP target cells
Drug: Fludarabine — Part of the non-myeloablative lymphocyte-depleting preparative regimen.
Drug: Cyclophosphamide — Part of the non-myeloablative lymphocyte-depleting preparative regimen.

SUMMARY:
Alkaline phosphatase (ALP) is a membrane-bound glycoprotein that catalyzes the hydrolysis of phosphates at alkaline pH values. As one of the earliest discovered oncofetal antigens, ALP has emerged as a significant biomarker for various malignant tumors, such as ovarian cancer, breast cancer, trophoblastic tumors, germ cell tumors, endometrial cancer, testicular tumors, cervical intraepithelial neoplasia, and gastrointestinal tumors.

DETAILED DESCRIPTION:
This is a single-center, open-label, study of CAR-T cells for the treatment of the recurrent/metastatic solid tumors patients who had failed standard therapy.

Objective:

To evaluate the safety and efficacy of CAR-T cells in the treatment of advanced solid tumors.

Eligibility:

Adults aging 18-70 with advanced solid tumors

Design:

1. Patients will undergo a comprehensive set of screening tests, including imaging procedures, evaluation of cardiac and pulmonary function, as well as a range of laboratory assessments.
2. After meeting the eligibility criteria and enrolling in the trial, patients will undergo leukapheresis for collection of autologous lymphocytes, which will be sent to manufacturing facilities.
3. Once cells have been manufactured, patients will then proceed to lymphodepleting chemotherapy followed by the infusion of ALPP CAR T-cells.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and sign the Informed of Consent Document. Be willing to follow the procedure and protocol of the clinical trial;
2. Age 18-70 (including boundary value), both male and female;
3. Expected life span is more than 3 months from the date of signing the informed consent;
4. ECOG score 0-1;
5. Metastatic or recurrent solid tumors confirmed by histopathology;
6. Refractory to standard treatment evaluated by radiological assessment;
7. Be able provide fresh or preserved tissue specimen;
8. At least 1 measurable lesion (according to RECIST 1.1);
9. ALPP expression positivity determined by IHC；
10. The organ marrow function of the subjects meets the following requirements:

    1. Marrow function：ANC≥ 1.5×109/L; PLT count≥ 75×109/L; HGB≥ 90 g/L;
    2. Coagulation function: Prothrombin Time (PT)≤ 1.5 times the Upper Limit of Normal (ULN), International Normalized Ratio (INR)≤ 1.5 times ULN, and Activated Partial Thromboplastin Time (APTT)≤ 1.5 times ULN;
    3. Liver function: ALT and AST≤ 2.5 times ULN (in cases of liver transfer/infiltration, ≤ 5.0 times ULN); Total Bilirubin (TBIL) ≤ 1.5 times ULN (with Gilbert's syndrome, <3×ULN);
    4. Renal function: Serum Creatinine (Cr)≤ 1.5 times ULN or Creatinine Clearance Rate (CrCl) ≥ 60ml/min;
    5. Cardiac function: Left Ventricular Ejection Fractions (LVEF)≥45%;
    6. Pulmonary function: Forced Expiratory Volume in the first second (FEV1) ≥ 50%.
11. Prior to the first dose, subjects must have recovered from toxic effects of previous treatment (CTCAE grade ≤ 1, with the exception of specific criteria such as "alopecia"), and the investigator determines that the corresponding adverse events do not pose a safety risk.
12. For male or female subjects of childbearing potential: from the time of signing the ICF until at least 24 weeks after the last dose, they must agree to practice abstinence or use effective contraceptive methods, including intrauterine devices, etc.

    Note: Women of childbearing potential who have undergone surgical sterilization (including hysterectomy, bilateral oophorectomy, or salpingectomy) or who have been postmenopausal for more than 24 months are considered to have no potential for pregnancy.
13. A suitable venous access for the necessary blood collection can be established, and there are no contraindications for leukapheresis.

Exclusion Criteria:

Inclusion criteria:

1. Be able to understand and sign the Informed of Consent Document. Be willing to follow the procedure and protocol of the clinical trial;
2. Age 18-70 (including boundary value), both male and female;
3. Expected life span is more than 3 months from the date of signing the informed consent;
4. ECOG score 0-1;
5. Metastatic or recurrent solid tumors confirmed by histopathology;
6. Refractory to standard treatment evaluated by radiological assessment;
7. Be able provide fresh or preserved tissue specimen;
8. At least 1 measurable lesion (according to RECIST 1.1);
9. ALPP expression positivity determined by IHC；
10. The organ marrow function of the subjects meets the following requirements:

    1. Marrow function：ANC≥ 1.5×109/L; PLT count≥ 75×109/L; HGB≥ 90 g/L;
    2. Coagulation function: Prothrombin Time (PT)≤ 1.5 times the Upper Limit of Normal (ULN), International Normalized Ratio (INR)≤ 1.5 times ULN, and Activated Partial Thromboplastin Time (APTT)≤ 1.5 times ULN;
    3. Liver function: ALT and AST≤ 2.5 times ULN (in cases of liver transfer/infiltration, ≤ 5.0 times ULN); Total Bilirubin (TBIL) ≤ 1.5 times ULN (with Gilbert's syndrome, <3×ULN);
    4. Renal function: Serum Creatinine (Cr)≤ 1.5 times ULN or Creatinine Clearance Rate (CrCl) ≥ 60ml/min;
    5. Cardiac function: Left Ventricular Ejection Fractions (LVEF)≥45%;
    6. Pulmonary function: Forced Expiratory Volume in the first second (FEV1) ≥ 50%.
11. Prior to the first dose, subjects must have recovered from toxic effects of previous treatment (CTCAE grade ≤ 1, with the exception of specific criteria such as "alopecia"), and the investigator determines that the corresponding adverse events do not pose a safety risk.
12. For male or female subjects of childbearing potential: from the time of signing the ICF until at least 24 weeks after the last dose, they must agree to practice abstinence or use effective contraceptive methods, including intrauterine devices, etc.

    Note: Women of childbearing potential who have undergone surgical sterilization (including hysterectomy, bilateral oophorectomy, or salpingectomy) or who have been postmenopausal for more than 24 months are considered to have no potential for pregnancy.
13. A suitable venous access for the necessary blood collection can be established, and there are no contraindications for leukapheresis.

Exclusion criteria:

1. Subjects with primary central nervous system (CNS) malignancies; subjects with CNS metastases who have failed local treatment; subjects without symptomatic brain metastases within 14 days before pretreatment, or with stable clinical symptoms and no requirement for corticosteroids or other treatment for brain metastases, may be included;
2. Prior history of malignancy with non-target indications within the past 5 years, with the exception of: adequately treated malignancies, with more than 5 years of stability and minimal risk of recurrence as judged by the investigator; and in situ carcinoma without evidence of recurrence after adequate treatment;
3. Subjects with any active autoimmune disease, history of autoimmune disease, or requiring systemic corticosteroids (≥10 mg/day prednisone equivalent) or immunosuppressive therapy, or syndromes (subjects with skin diseases that do not require systemic treatment or have resolved childhood asthma/allergies without any intervention as an adult; subjects with stable thyroid hormone replacement therapy for autoimmune hypothyroidism may be included);
4. History of immunodeficiency, including positive HIV testing or other acquired or congenital immunodeficiency diseases;
5. History of hereditary or acquired bleeding disorders;
6. Presence of cardiovascular clinical conditions or symptoms, including: a. History of thromboembolic events ≥ grade 3 in the past 6 months, or currently receiving thrombolytic or anticoagulant therapy due to high thrombotic risk; b. Chronic heart failure with reduced ejection fraction (NYHA class ≥ II); c. History of unstable angina; d. Myocardial infarction in the past 6 months; e. Clinically significant malignant arrhythmias (excluding atrial fibrillation, paroxysmal supraventricular tachycardia); f. Clinically significant QTcF prolongation (QTcF > 450 ms for males, QTcF > 470 ms for females, derived from Fridericia's formula); g. Poorly controlled hypertension.
7. Presence of active infection (fever due to tumor growth may be included as judged by the investigator);
8. Active pulmonary tuberculosis detected by history or CT scan, or history of active pulmonary tuberculosis within the past 1 year before inclusion, or history of active pulmonary tuberculosis more than 1 year ago without proper treatment;
9. Patients with active hepatitis B or hepatitis C virus infection (active hepatitis B defined as hepatitis B virus deoxyribonucleic acid (HBV-DNA) > the lower limit of detection; active hepatitis C defined as hepatitis C virus ribonucleic acid (HCV-RNA) > the lower limit of detection) or positive syphilis serology;
10. Pregnant or lactating women, or subjects with a positive blood pregnancy test;
11. Serious surgery or major trauma within 28 days before lymphodepletion;
12. Vaccination with live or attenuated vaccines within 28 days before Lymphodepletion;
13. Systemic corticosteroids (excluding inhaled therapy, topical treatment, or physiological replacement therapy) or other immunosuppressive treatments within 14 days before lymphodepletion;
14. Receiving any investigational drug or participating in another clinical study within 28 days before lymphodepletion (except for subjects participating in observational, non-interventional clinical studies, or in the survival follow-up period of an interventional clinical study);
15. Refractory or persistent seizures, significant pleural or abdominal effusions, active gastrointestinal bleeding, or subjects judged by the investigator to be at high risk of significant bleeding due to tumor necrosis;
16. Concomitant severe organic or psychiatric diseases;
17. Prior history of allogeneic bone marrow or solid organ transplantation, or renal replacement therapy;
18. Under the investigator's judgment, subjects with uncontrollable tumor-related pain or compression symptoms due to a large tumor burden that requires palliative treatment or radiation therapy should have completed treatment before entering the study;
19. History of substance abuse, or alcohol or drug abuse;
20. Prior cellular therapy (TCR-T, CAR-T, TIL, etc);
21. Prior severe allergic reaction to any drug or its components in this trial;
22. Subjects whose condition is judged by the investigator to be unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity or Maximum Tolerated Dose (MTD) | Day 28 post-initial ALPP CAR-T infusion
  Dose Limiting Toxicity (DLT) is defined as patients with the adverse event (AE) or laboratory abnormality assessed by the principal investigator (PI). These should be possibly related to ALPP CAR-T cell therapy, and should be unrelated to the disease itself, disease progression, concomitant diseases or concomitant medication. The MTD is the highest dose at which no more than one out of six patients experiences DLT, or the highest dose level tested if no DLTs are observed across all dose levels.
Overall response rate | Day 0 - Day 730
  The efficacy of ALPP CAR-T is assessed by the objective response rate (ORR) according to RECIST 1.1 and iRECIST. ORR is defined as patients who have achieved either a partial response (PR) or a complete response (CR).
Treatment-related adverse events as assessed by CTCAE v5.0 | Day 0 - Day 730
  The type, incidence and severity of adverse events include clinically significant post-treatment abnormal laboratory examination results, abnormal physical examination and blood examination results, bone marrow examination results, etc. Clinical and laboratory AEs will be classified according to the National Cancer Institute general terminology standard for adverse events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Duration of response | Day 0 - Day 730
  The efficacy of ALPP CAR-T will be assessed by duration of response (DOR). The DOR refers to the length of time from the first appearance of a treatment response to the first occurrence of progressive disease or recurrence.
Progression free survival | Day 0 - Day 730
  The efficacy of ALPP CAR-T will be assessed by progression free survival (PFS). The PFS refers to the time from treatment to progressive disease or death for any reason.
Overall survival | Day 0 - Day 730
  The efficacy of ALPP CAR-T will be assessed by overall survival (OS). The OS refers to the time from treatment to death.
Expansion and persistence of ALPP CAR-T cells in peripheral blood or serous effusion (if present) | Day 0 - Day 730
  Blood and serous effusion (if present) samples were collected to measure persistence of infused ALPP CAR-T using polymerase chain reaction of a vector specific sequence in deoxyribonucleic acid (DNA) extracted from peripheral blood mononuclear cell (PBMC).
Cell cytokine levels and tumor biomarkers in peripheral blood and serous effusion (if present) | Day 0 - Day 730
  Blood samples and serous effusion (if present) were collected to measure cytokines IL-6, TNF-α, IL-8, IFN-γ, C-reactive protein (CRP), as well as ALPP concentration, Alpha-fetoprotein (AFP), Human chorionic gonadotropin (hCG), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Qingzhu Jia, M.D., Principal Investigator — Xinqiao Hospital
Locations (1):
- Department of Hematology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No